CLINICAL TRIAL: NCT06087302
Title: Effectiveness of Child-Parent Relationship Therapy (CPRT) for Management of Psychological Distress and Family Functioning Among Parents of Children Exposed to Trauma
Brief Title: Effectiveness of Child-Parent Relationship Therapy (CPRT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Tayyaba Hanif, Ph.D. scholar, Fatima Jinnah Women University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: FJWU/EC/2023/60
Record Dates: First submitted 2023-10-03; First posted 2023-10-17 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Behavior Disorders in Children
Keywords: Child Parent relationship therapy; Family functioning,; Psychological distress; child exposed to Trauma; disruptive behavior
MeSH Terms: conditions — Child Behavior Disorders; Problem Behavior

STUDY DESIGN:
Intervention Model Description: Child-Parent Relationship Therapy (CPRT) is a play-established therapy process for young children, aged between 3-10, who have attachment issues, and behavioral, social, or emotional issues. It is based on ten weekly, two-hour group sessions for a group of 5-8 members in the group. Learning skills, receiving feedback on skill practice, and connecting with other parents for support are all critical components of the CPRT program. Parents learn skills and prepare for future play sessions with their children during sessions 1-3. Parents practice their new skills with their children in weeks 4-10, while the therapist provides feedback in a small group setting.
Who Masked: Participant, Investigator
Masking Description: there would be two groups intervention group and a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): the control group wouldnot receive the CPRT for caregivers/parents
- CPRT intervention group (Experimental): intervention group would receive the CPRT for caregivers/parents
  Interventions: Behavioral: child-Parent Relationship Therapy (CPRT)

INTERVENTIONS:
Behavioral: child-Parent Relationship Therapy (CPRT) — The Child Parent Relationship Therapy (CPRT) is an evidence-based intervention program that trains parents/caretakers to help their children with social, emotional, attachment, and behavioral difficulties
  Arms: CPRT intervention group

SUMMARY:
Exposure to trauma during childhood contributes to behavioral and attachment difficulties in children. The current research study will be conducted on the effectiveness of child-parent relationship therapy (CPRT) on psychological distress and family functioning among parents of children exposed to trauma. The CPRT is an evidence-based intervention parenting program that gives training to the parents, to help children who have social, emotional, attachment, and behavioral difficulties. A CPRT would train parents with the principles of CCPT and provide them with the ability to support their children. A randomized controlled trial will validate the effect of CPRT on family functioning, and parental psychological distress among parents of children exposed to trauma. It will be an interventional-based study on CPRT with a pre-posttest experimental design. The current study would be conducted in Islamabad and Rawalpindi, after obtaining permission from the appropriate authorities, for collecting data from the educated mothers/caretakers as a research sample. There would be inclusive and exclusive selection criteria for the sample. A study will be conducted in four ways, firstly, the need assessment will be conducted with phenomenological research design from selected educated mothers/caretakers on the KAP model (knowledge, attitudes, and practices) categories about the CPRT, and psychological distress on family functioning among parents of children exposed to trauma. In phase two, the pilot study will be conducted to assess the accuracy of measures for the sample and the effectiveness of CPRT. In phase three, a cross-sectional survey would measure the study variables. The fourth phase will be the intervention phase for validation of CPRT therapeutic techniques in the Pakistani population a randomized controlled trial design will be applied to analyze the effect of CPRT on study variables in the next phase (main study). The measures Child-Parent Relationship Scale, depression, anxiety, and stress scale, family assessment device, and disruptive behavior through Children's Behavior Questionnaire (very short form) parental-version will be used to collection the data from study participants. The Child and Adolescent Trauma Screen would be used as a screening inventory. The CPRT intervention therapeutic sessions will continue based on the inclusive and exclusive selection criteria. The data will be evaluated through SPSS (latest version).

DETAILED DESCRIPTION:
Nature of Study The proposed study is primary in nature. A primary data collection is intended for the current study, which would gather information from parents of children exposed to trauma Study Design The proposed research design, the current study would be centered on a mixed research design to measure study objectives. The objectives are based on the exploratory qualitative design and cross-sectional experimental research design. The study would adopt the mixed methodology (exploratory research design, cross-sectional research design) and randomized controlled experimental method (in terms of pre and post-intervention effects).

The child-parent relationship (in the context of closeness and conflict) would predict the primary outcome of family functioning (in the context of Warmth, Communication, Support conflicts, and worries) and psychological distress (in the context of depression, anxiety, stress). The secondary outcome would be the child's behavior (in the context of internalized symptoms of Grief/ Loss and anxiety/Mood). Child Parent-relationship therapy would be used for implementation to study the level of family functioning and psychological distress. CPRT will introduce special play time to the parent for the children exposed to trauma and will study the level of internalized symptoms of the child's behavior. The current study would find out the effectiveness of CPRT on child-parent relationships, parental psychological distress in family functioning, and parents of children exposed to trauma in twin cities of Pakistan.

During study one, the exploratory research design will be used to collect the data from the selected sample on knowledge, attitudes, and practices categories about the parent-child relationship, and psychological distress on family functioning among parents of children exposed to trauma. phase one is a pilot study. During phase two, a baseline survey will be conducted to see the association between the study variables and differences between the demographic characteristics of the sample.

During phase three Randomized controlled trial (RCT), will be used for: a) Mean scores validation of Child-parent relationship therapeutic techniques in the Pakistani family functioning. b) The parents of children exposed to trauma who receive intensive child-parent relationship training attain a comparison of level of psychological distress mean scores of DASS between the group compared with non-treatment comparison group parents of children exposed to trauma c) The Comparison between the mean scores of the Children's Behavior Questionnaire (concise form) parental version of children's disruptive behavior and significant difference between the pre-testing and post-testing. d) comparison between within a group mean scores of child-parent relationship scale in post-testing. e) Differences in mean scores between the experimental group's pre- and post-testing results and, f) Statistical mean score based on post-testing assessment results, statistical mean score differences will be evaluated between experimental and control groups.

Sample Research participants would be selected initially with snowball sampling techniques and later with purposive sampling. Research participants would be recruited including educated mothers (minimum qualification would be graduation 14 years of qualification) from twin cities (Rawalpindi and Islamabad) of Pakistan. The demographic characteristics of the sample would be, family system (joint family, and nuclear family system) , marital status(married, widow, separated/divorced), and monthly income and age. Additional inclusive sample criteria also include the parents of children exposed to traumatic experiences, child abuse, bullying, fighting, accidents, traumatized grief, and parents' separation. Exclusive Sample criteria will not include uneducated parents, domestic violence child sexual abuse, natural disasters, traumatic events that caused physical disabilities, war, terrorism victims, and families who would be taking any psychotherapy or training for the management of psychological distress and child disruptive behavior. Each potential parent would be screened briefly through screening inventories for all phases of the current study. Before every interview, the researcher would be clear the objectives of the current study. The ethical considerations would be considered for selected research participants for all phases.

Phase-I research participants would be fifteen to twenty-five educated mothers' target. The data will be collected through semi-structured interviews till the time of saturation. Phase-II research participants would be calculated through Raosoft. Phase III there would be n=x research participants finalized for the experimental group after the screening and would meet the inclusion criteria. The experimental group would be divided into 8 groups. There would be 8 research participants in each group as the requirement of the CPRT protocol. A randomization process ensures that all research participants have the same demographic characteristics in intervention and control groups. The children's age should be between 3-10 years as it is a basic criterion of child-parent relationships. The pre-testing session would be conducted before the intervention phase. The post-testing session would be conducted after the intervention phase.

Furthermore, it is not always possible to meet randomization requirements in educational research studies, thus an extensive reliance on numbers may not be an adequate representation. Available resources, time constraints, and the number of volunteers that would be willing to participate in a study govern sample size in research, especially in educational research. Therefore, approximately 30-60 parents of children exposed to trauma would be randomly split into interventional and control groups after initial assessment.

Measures According to all phases of the current study, different measurements will be used to meet the objectives. A study will be conducted in three ways, firstly, the need assessment will be conducted with exploratory research design from selected educated mothers/caretakers on knowledge, attitudes, and practices categories about the relationship between parents and children, psychological stress, family functioning of parents of traumatized children experiences psychological distress. For need assessment, therefore semi-structured interview protocol will be developed according to the categories identified from the literature. A cross-sectional survey will be conducted in phase two to see the relationship between the study variables. To validate CPRT therapeutic techniques in the Pakistani population, a randomized controlled trial design will be used to examine the impact of CPRT on study variables in the next phase (main study). The measures of the Child-Parent Relationship Scale, depression, anxiety, stress scale, family assessment device, The child and adolescent Trauma Screen, and disruptive behavior through the child and adolescent Behavior inventory parental version.

ELIGIBILITY:
Inclusion Criteria:

1. qualification would be graduation minimum and above
2. location: from Pakistan's twin cities (Rawalpindi and Islamabad). 3. the parents of children exposed to traumatic experiences

   * child abuse (physical abuse, yelling, Psychological Abuse)
   * bullying, (witness of bullying, verbal bullying, physical bullying)
   * fighting, (street fighting. witness of fighting)
   * traumatized grief, (death of a loved one)
   * Robbery and
   * parents' separation.

Exclusion Criteria: Exclusive Sample criteria

* uneducated parents, (less then graduation)
* domestic violence
* child sexual abuse,
* natural disasters,
* traumatic events that caused physical disabilities,
* war,
* terrorism victims, and
* families who would be taking any psychotherapy or training to manage psychological distress and child disruptive behavior.

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — mothers of children between 3-10 years would be part of the study
Enrollment: 60 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-09 (Estimated)

PRIMARY OUTCOMES:
Child Parent Relationship Scale | 10-15 minutes
  it consists of fifteen items about the child and the parent's relationship with it. Likert weighed the fifteen items on a 5-point scale, and CPRS can be summarized by groups of objects that most closely correspond to the discrepancy and closeness.
Depression Anxiety Stress Scale-42 | 5-10 minutes
  it is based on measurements rather than categorical concepts of mental distress, and scores emphasize symptoms are experienced, not diagnostic thresholds. it has been unable to use a child's scale for 12 years, The three symptom clusters are as follows: Depression: Illegal problems, despair, life assessment, vertical, pride, interest/involvement, and tribe/involvement, Anxiety: Herbal arousal, skeletal muscle effects, conditional warnings, fear of anxiety. Stress: Chronic non-special Here, the complexity is comfortable, nervous, easily frustrated/excited, sensitive/impatient beyond.
Family Assessment Device | 10-15 minutes
  measures structural, organizational, and transactional factors within families. A total of six scales are used to measure the six dimensions of the MMFF - affective involvement, affective responsiveness, behavioral control, communication, problem solving, and roles - as well as a seventh measure measuring general family functioning

SECONDARY OUTCOMES:
Child and adolescent Behavior Inventory | 5-10 minutes
  A children's behavior questionnaire was used to assess the child's behavior. There were 75 items with 3-point Likert scale and evaluation for last 6 months.. it is suitable for the age range of the child between 6-17 years.

OTHER OUTCOMES:
Child and Adolescent Trauma Screen-Caregiver | 5-10 minutes
  The questionnaire is indeed a screening tool designed to assess potentially traumatic events and posttraumatic stress symptoms (PTSS) in children and adolescents. It is based on the DSM-5 criteria for PTSD. The CATS questionnaire typically consists of questions related to traumatic events and symptoms associated with PTSD. According to the DSM-5, (2013) the CATS measures potentially traumatic experiences and posttraumatic stress symptoms (PTSS). age 3-17 y

CONTACTS AND LOCATIONS:
Locations (1):
- Tayyaba Hanif, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No